CLINICAL TRIAL: NCT06531577
Title: Influence of Atmospheric Pressure on Patients Presenting to the Emergency Department With Epistaxis
Brief Title: Atmospheric Pressure and Epistaxis Relationship
Status: Recruiting | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: Ankara Etlik City Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: atmospheric pressure
Record Dates: First submitted 2024-07-17; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Atmospheric Pressure; Adverse Effect; Epistaxis Nosebleed
Keywords: atmospheric pressure; epistaxis; blood pressure
MeSH Terms: conditions — Epistaxis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- epistaxis group: patients presenting to emergency department with epistaxis

SUMMARY:
In this study, investigators aim to understand the relationship between changes in atmospheric pressure and blood pressure, and to investigate whether these changes have an impact on the etiology of epistaxis.

DETAILED DESCRIPTION:
This study aims to investigate the potential effects of changes in atmospheric pressure on epistaxis and, if such effects exist, to review treatment adjustments based on weather forecasts for hypertensive patients to prevent potential hypertensive emergencies and enhance patient comfort. This research poses no risk to patients and is purely observational and clinical in nature.

The study will be conducted prospectively over a period of 6 months at the Emergency Department of Ankara Etlik City Hospital, focusing on patients presenting with epistaxis.After initial evaluation upon presentation to the emergency department, patients will undergo routine emergency department monitoring for epistaxis, including physical examination, vital sign monitoring, evaluation of coagulation parameters, and hemoglobin levels. Apart from routine tests, no additional invasive or non-invasive procedures will be performed by us.

Data obtained from patients and daily atmospheric pressure parameters will be evaluated and analyzed.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18 and above Presenting to the emergency department with complaints of epistaxis, whether active or resolved.

Willing volunteers consenting to participate in the study. Residing in central districts of Ankara

Exclusion Criteria:

Patients under the age of 18. Pregnant individuals. Those with a history of maxillofacial surgery. Patients reporting a history of trauma at the time of admission. Patients stating they are from a city other than Ankara.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients over the age of 18 presenting to emergency department with epistaxis
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
epistaxis | 24 hours
  number of the patients with epistaxis will be evaluated accoridng to atmospheric preesure and wheather conditions on daily basis

CONTACTS AND LOCATIONS:
Overall Officials: gulsen akcay, ass. prof., Study Director — ass. prof. of organization
Locations (1):
- Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jelavic B, Majstorovic Z, Kordic M, Leventic M, Grgic MV, Baudoin T. Idiopathic epistaxis and meteorological factors: case-control study. B-ENT. 2015;11(4):267-73. PMID 26891538
- [Background] Min SJ, Kang H, Kim KS, Min HJ. Minimal temperature, mean wind speed, and mean relative humidity are associated with spontaneous epistaxis in Seoul, Korea. Auris Nasus Larynx. 2021 Feb;48(1):98-103. doi: 10.1016/j.anl.2020.07.012. Epub 2020 Jul 25. PMID 32718810